CLINICAL TRIAL: NCT02150655
Title: Pilot Study Investigating Bacteria (Microbiota), Their By-products (Metabolome) and Environmental Toxins in Relation to Reproductive Health in Rwandan Women.
Brief Title: Study of the Microbiota, Metabolome, and Environmental Toxins in Relation to Reproductive Health in Rwandan Women
Acronym: RVMM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Gregor Reid, Director, Canadian R&D Centre for Probiotics, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 102886
Record Dates: First submitted 2013-07-04; First posted 2014-05-30 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Vulvovaginal Candidiasis; Bacterial Vaginosis
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Vaginosis, Bacterial | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14 oral capsules
  Interventions: Biological: Lactobacillus GR-1 and Lactobacillus RC-14 oral capsules
- Placebo (Placebo Comparator): Sugar pill
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Lactobacillus GR-1 and Lactobacillus RC-14 oral capsules
  Arms: Probiotic
Biological: Placebo
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The overall objective of this clinical pilot study is to determine at a random sampling time, the vaginal microbiome and metabolome of pregnant women, and to see if infection (bacterial vaginosis, vulvovaginal candidiasis, malaria) and exposure to environmental toxins affects could alter pregnancy and conception outcomes. It is hypothesized that infection and toxins will alter the vaginal microbiome and metabolome, increasing the risk of preterm labour and infertility in Rwandan women. In a sub-group of subjects, a preliminary assessment of the ability of orally administered probiotic lactobacilli to restore the vaginal microbiota to a healthy state and lower environmental toxins will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18 and 55.

Exclusion Criteria:

* *Current infection of gonorrhoea, *Chlamydia, genital warts, *active genital herpes lesions, *active syphilis; *urinary tract infection including pyelonephritis (an ascending urinary tract infection); *receiving drug therapy that may affect the vaginal flora; *had unprotected sexual intercourse (vaginal or oral) within the past 48 hours; *have used a vaginal douche, genital deodorant, or genital wipe products in the past 48 hours; *have taken any 'acidophilus' 'bifidobacteria' or probiotic health food supplements in the past 48 hours; *are menstruating at time of clinical visit.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
maintenance of healthy vaginal microbiota | 1 month
  The change in relative abundance of healthy lactobacilli and species associated with bacterial vaginosis after one month probiotic intervention will be assessed using 16S rRNA gene sequencing.

SECONDARY OUTCOMES:
Reduction of environmental toxins in blood by lactobacilli | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Dr Reid, PhD, Principal Investigator — Western University, Canada
Locations (1):
- Nyamata District Hospital, Nyamata, East Province, Rwanda

REFERENCES:
- [Derived] McMillan A, Rulisa S, Gloor GB, Macklaim JM, Sumarah M, Reid G. Pilot assessment of probiotics for pregnant women in Rwanda. PLoS One. 2018 Jun 18;13(6):e0195081. doi: 10.1371/journal.pone.0195081. eCollection 2018. PMID 29912913